CLINICAL TRIAL: NCT07236593
Title: Remnant Preservation in Anterior Cruciate Ligament Reconstruction: Does Stump Suturing Reduce the Risk of Tibial Tunnel Widening? A CT-Based Study
Brief Title: Remnant Preservation and Tibial Tunnel Widening After ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed El-Desouky, Associate Professor of Orthopedic surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-473-2021
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stump-Suturing ACL Reconstruction (Experimental)
  Interventions: Procedure: Stump-Suturing ACL Reconstruction
- Stump-Resection ACL Reconstruction (Active Comparator)
  Interventions: Procedure: Stump-Resection ACL Reconstruction

INTERVENTIONS:
Procedure: Stump-Suturing ACL Reconstruction — Patients in this group undergo arthroscopic ACL reconstruction with preservation and suturing of the native ACL remnant (stump) around the graft. The technique aims to enhance graft revascularization and biological healing, potentially reducing tibial tunnel widening.
  Arms: Stump-Suturing ACL Reconstruction
Procedure: Stump-Resection ACL Reconstruction — Patients in this group undergo standard arthroscopic ACL reconstruction with complete resection of the ACL remnant (stump) prior to graft placement. This represents the conventional surgical approach for ACL reconstruction.
  Arms: Stump-Resection ACL Reconstruction

SUMMARY:
Anterior Cruciate Ligament (ACL) reconstruction is one of the most commonly performed orthopedic procedures. Tibial tunnel widening is a recognized postoperative complication that may affect graft stability and long-term outcomes. Recent studies have suggested that preserving the ACL remnant may improve biological healing and reduce tunnel widening, but the evidence remains inconclusive.

This prospective randomized study aims to evaluate whether remnant (stump) preservation and suturing during ACL reconstruction can reduce the risk of tibial tunnel widening compared with the conventional stump-resection technique.

A total of 190 patients with recent ACL tears (<6 months) were randomly assigned into two equal groups: Group A underwent arthroscopic ACL reconstruction with remnant suturing, while Group B underwent standard reconstruction with stump resection. All patients were followed for 12 months postoperatively with serial CT evaluations to assess tunnel diameters and positioning.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Acute ACL injury (<6 months)
* Medically fit for surgery

Exclusion Criteria:

* Age <18 or >45 years
* Old or chronic ACL injuries (>6 months)
* Multi-ligamentous knee injuries
* Failed previous ACL reconstruction
* Associated mal-alignment deformities
* Absence of identifiable ACL stump

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Rate of Tibial Tunnel Enlargement | 12 months postoperatively

SECONDARY OUTCOMES:
Percentage of Tibial Tunnel Enlargement | 12 months
Tibial Tunnel Positioning (X & Y coordinates) | 2 Weeks
Femoral Tunnel Diameter Change | 12 months
Femoral Tunnel Positioning (X & Y coordinates) | 2 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt